CLINICAL TRIAL: NCT05004935
Title: Analysis of Electromyography Activation Trunk Muscles and the Effect of Beetroot Juice Intake on the Results in Strength Exercises: Lateral Medicine Ball Throw and Sled Pushing
Brief Title: The Effect of Beetroot Juice on Plasma Trimethylamine N-oxide Concentration
Acronym: BRJ_TMAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Robert Olek, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RMPN2021/JJ
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nitrates

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beetroot juice (Experimental): single intake of beetroot juice containing 800mg nitrates
  Interventions: Dietary Supplement: beetroot juice
- nitrates (Active Comparator): single intake of 800mg nitrates (NaNO3)
  Interventions: Other: nitrate

INTERVENTIONS:
Dietary Supplement: beetroot juice — single intake of beetroot juice containing 800mg nitrates
  Other Names: 140 ml of Beet It juice
  Arms: beetroot juice
Other: nitrate — single intake of 800mg nitrates
  Other Names: NaNO3
  Arms: nitrates

SUMMARY:
The primary aim of the current study is to determine the effect of beetroot juice consumption on plasma trimethylamine N-oxide concentration.

A secondary aims: exploring the effect of circulating trimethylamine N-oxide modification on plasma total antioxidant status, and measurement of changes in the skin nicotinamide-adenine dinucleotide reduced form (NADH) content during transient ischemia and reperfusion.

DETAILED DESCRIPTION:
In a random order subjects will consume beetroot juice (140ml), or equimolar nitrates (NaNO3). Antecubital vein blood samples will be taken at the beginning, and every hour for 4 hours following consumption.

Plasma trimethylamine N-oxide, total antioxidant status, and nitrite/nitrate concentrations will be determined.

Using Flow Mediated Skin Fluorescence skin NADH content determined during controlled ischemia triggered by total occlusion of the brachial artery by the brachial blood pressure cuff and during reperfusion after deflation of the blood pressure cuff 2 and 4 hours following consumption.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers

Exclusion Criteria:

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The effect of beetroot juice consumption on plasma trimethylamine N-oxide concentration | 4 hours
  Determination of plasma trimethylamine N-oxide concentration following the beetroot juice consumption using ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS) method.

SECONDARY OUTCOMES:
The effect of circulating trimethylamine N-oxide modification on plasma total antioxidant status | 4 hours
  Determination of plasma total antioxidant status following the beetroot juice consumption using commercially available kit.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olek, PhD, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Akademia Wychowania Fizycznego, Poznan, Poland

REFERENCES:
- [Derived] Jurga J, Samborowska E, Zielinski J, Olek RA. Effects of Acute Beetroot Juice and Sodium Nitrate on Selected Blood Metabolites and Response to Transient Ischemia: A Crossover Randomized Clinical Trial. J Nutr. 2024 Feb;154(2):491-497. doi: 10.1016/j.tjnut.2023.12.018. Epub 2023 Dec 16. PMID 38110180